CLINICAL TRIAL: NCT02959775
Title: Immunogenicity and Safety of High-dose Hepatitis B Vaccine Among Drug Users: a Randomized, Controlled Trial
Brief Title: Immunogenicity of Hepatitis B Vaccination Among Drug Users
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanxi Medical University (Other)
Collaborators: Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Principal Investigator, Suping Wang, Professor, Shanxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2012ZX10002001003004002
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Results first posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2021-12

CONDITIONS: Hepatitis B Vaccination
Keywords: Hepatitis B vaccination; Immunogenicity; Randomized controlled trial; Drug abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 60 µg dose hepatitis B vaccine (Experimental): Receive three intramuscular injections of 60 µg recombinant hepatitis B vaccine at months 0, 1 and 6
  Interventions: Biological: 60 µg dose hepatitis B vaccine
- 20 µg dose hepatitis B vaccine (Experimental): Receive three intramuscular injections of 20 µg recombinant hepatitis B vaccine at months 0, 1 and 6
  Interventions: Biological: 20 µg dose hepatitis B vaccine
- Control (No Intervention): Receive no vaccination during the study period

INTERVENTIONS:
Biological: 60 µg dose hepatitis B vaccine — three-dose, 60 µg per dose
  Arms: 60 µg dose hepatitis B vaccine
Biological: 20 µg dose hepatitis B vaccine — three-dose, 20 µg per dose
  Arms: 20 µg dose hepatitis B vaccine

SUMMARY:
Uptake, adherence, and completion of vaccination among drug users were low, and their immune function and immune response to hepatitis B vaccination were also suboptimal, indicating that the current practice of hepatitis B vaccination can't protect drug users from HBV infection.

This is a randomized, open-label, blank-controlled trial, conducted among drug users with drug rehabilitation. This study will compare the immunogenicity and safety of three intramuscular 20µg and 60µg recombinant hepatitis B vaccines at months 0, 1, and 6 among drug users

DETAILED DESCRIPTION:
Comparison of 2 vaccination strategy against Hepatitis B in Drug Users

Intervention:

Arm 1 : Receive three intramuscular injections of 60 µg recombinant hepatitis B vaccine at months 0, 1 and 6;

Arm 2 : Receive three intramuscular injections of 20 µg recombinant hepatitis B vaccine at months 0, 1 and 6;

Arm 3 : Receive no vaccination during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years at the enrolment
* current illicit drug users before drug rehabilitation
* negative for hepatitis B surface antigen (HBsAg) and hepatitis B surface antibody (anti-HBs) at enrollment
* having spent acute physiological detoxification phase

Exclusion Criteria:

* any intolerance or allergy to any component of the vaccine
* ongoing opportunistic infection
* liver disease
* hemopathy
* cancer
* unexplained fever in the last week before the recruiting

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suping Wang, Principal Investigator — Shanxi Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Feng Y, Shi J, Gao L, Yao T, Feng D, Luo D, Li Z, Zhang Y, Wang F, Cui F, Li L, Liang X, Wang S. Immunogenicity and safety of high-dose hepatitis B vaccine among drug users: A randomized, open-labeled, blank-controlled trial. Hum Vaccin Immunother. 2017 Jun 3;13(6):1-7. doi: 10.1080/21645515.2017.1283082. Epub 2017 Mar 16. PMID 28301282

RESULTS

PARTICIPANT FLOW:
Groups:
- IM20 Group: Participants received 3 intramuscular injections of 20 μg recombinant hepatitis B vaccine at months 0, 1 and 6.
- IM60 Group: Participants received 3 intramuscular injections of 60 μg recombinant hepatitis B vaccine at months 0, 1 and 6.
- Blank Control Group: Participants received no intervention.
Period: Overall Study
Arm/Group | IM20 Group | IM60 Group | Blank Control Group
Started | 160 | 160 | 160
Completed | 133 | 133 | 124
Not Completed | 27 | 27 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IM20 Group | IM60 Group | Blank Control Group | Total
Number analyzed (Participants) | 160 | 160 | 160 | 480
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (8.7) | 36.4 (8.6) | 36.7 (8.3) | 36.7 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 160 | 160 | 160 | 480
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han ethnicity | 158 | 158 | 158 | 474
  minority ethnicity | 2 | 2 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  China: Urban | 67 | 62 | 69 | 198
  China: Rural | 93 | 98 | 91 | 282

OUTCOME MEASURES:

1. Primary Outcome: Number and Rate of Participants With Anti-HBs Seroconversion at Month 7
Description: The measurements of anti-HBs antibodies were determined quantitatively by CMIA（Chemiluminescent Microparticle Immunoassay）. The accepted protective serum anti-HBs level was ≥10 mIU/ml.
Time Frame: Month 7
Population: Exclusion of participants who did not received/competed vaccine or left the centers.150, 149 and 151 patients in the IM20, IM60 and blank control groups completed the followed-up at months 7 .
Measure: Count of Participants; unit: Participants
Arm/Group | IM20 Group | IM60 Group | Blank Control Group
Number analyzed (Participants) | 150 | 149 | 151
Participants | 142 | 138 | 0

2. Secondary Outcome: Anti-HBs Concentration at Month 7
Description: The measurements of anti-HBs antibodies were determined quantitatively by CMIA（Chemiluminescent Microparticle Immunoassay）.
Time Frame: Month 7
Measure: Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | IM20 Group | IM60 Group | Blank Control Group
Number analyzed (Participants) | 150 | 149 | 151
mIU/mL | 909.6 [671.8 to 1147.5] | 2022.5 [1379.8 to 2665.1] | 0.3 [0.2 to 0.5]

3. Secondary Outcome: Anti-HBs Concentration at Month 12
Description: as for outcome 2
Time Frame: Month 12
Population: 133, 133 and 124 patients in the IM20, IM60 and blank control groups completed the followed-up at months 12 .
Measure: Mean (95% Confidence Interval); unit: mIU/mL
Groups:
- Control: Participants received no intervention.
Arm/Group | IM20 Group | IM60 Group | Control
Number analyzed (Participants) | 133 | 133 | 124
mIU/mL | 470.5 [268.3 to 672.8] | 676.7 [458.8 to 894.6] | 0.3 [0.2 to 0.6]

4. Secondary Outcome: Number and Rate of Participants With Anti-HBs Seroconversion at Month 12
Description: as for outcome 1
Time Frame: Month 12
Population: 133, 133 and 124 patients in the IM20, IM60 and blank control groups completed the followed-up at months 12.
Measure: Count of Participants; unit: Participants
Arm/Group | IM20 Group | IM60 Group | Blank Control Group
Number analyzed (Participants) | 133 | 133 | 124
Participants | 119 | 122 | 0

5. Secondary Outcome: Occurrence of Adverse Events After Vaccination
Description: Occurrence of adverse reactions within 7 days after vaccination with the hepatitis B
Time Frame: Within 7 days after the vaccination, at Month 0, 1, and 6
Population: 158 participants in the IM20 group and 156 in the IM60 group received the ﬁrst injection. The blank control group was not vaccinated with hepatitis B vaccine, so adverse reactions of hepatitis B vaccine were not collected and analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | IM20 Group | IM60 Group
Number analyzed (Participants) | 158 | 156
Participants | 14 | 13

6. Secondary Outcome: Occurrence of Adverse Events After Vaccination
Description: Occurrence of adverse reactions within 28 days after vaccination with the hepatitis B
Time Frame: Within 28 days after the vaccination, at Month 0, 1, and 6
Population: The blank control group was not vaccinated with hepatitis B vaccine, so adverse reactions of hepatitis B vaccine were not collected and analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | IM20 Group | IM60 Group
Number analyzed (Participants) | 158 | 156
Participants | 2 | 2

7. Secondary Outcome: Serious Adverse Events (SAE) Occurred During Month 12
Time Frame: Month 0-12
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | IM20 Group | IM60 Group
Number analyzed (Participants) | 133 | 133
Participants | 0 | 0

8. Other Pre Specified Outcome: Number and Rate of Participants With Anti-HBs High-level Response at Month 7
Description: The measurements of anti-HBs antibodies were determined quantitatively by CMIA. and anti-HBs concentrations ≥100 mIU/ml were high-level response.
Time Frame: Month 7
Measure: Count of Participants; unit: Participants
Arm/Group | IM20 Group | IM60 Group | Blank Control Group
Number analyzed (Participants) | 150 | 149 | 151
Participants | 111 | 116 | 0

9. Other Pre Specified Outcome: Number and Rate of Participants With Anti-HBs High-level Response at Month 12
Description: as for outcome 8
Time Frame: Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | IM20 Group | IM60 Group | Blank Control Group
Number analyzed (Participants) | 133 | 133 | 124
Participants | 73 | 91 | 0

10. Other Pre Specified Outcome: Anti-HBs Concentration at Month 6 Before the Third Injection
Description: Anti-HBs concentration at month 6 before the third injection by CMIA
Time Frame: Month 6 before the third injection
Population: 155 and 150 patients in the IM20 and IM60 groups completed the followed-up at months 6 before the third injection.
Measure: Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | IM20 Group | IM60 Group | Blank Control Group
Number analyzed (Participants) | 155 | 150 | 151
mIU/mL | 126.3 [49.5 to 203.2] | 524.5 [109.3 to 939.7] | 0.3 [0.2 to 0.5]

11. Other Pre Specified Outcome: Number and Rate of Participants With Anti-HBs Seroconversion at Month 6 Before the Third Injection
Description: The measurements of anti-HBs antibodies were determined quantitatively by CMIA. The accepted protective serum anti-HBs level was ≥10 mIU/ml.
Time Frame: Month 6 before the third injection
Measure: Count of Participants; unit: Participants
Arm/Group | IM20 Group | IM60 Group | Blank Control Group
Number analyzed (Participants) | 155 | 150 | 151
Participants | 98 | 109 | 0

12. Other Pre Specified Outcome: Number and Rate of Participants With Anti-HBs High-level Response at Month 6 Before the Third Injection
Description: as for outcome 8
Time Frame: Month 6 before the third injection
Measure: Count of Participants; unit: Participants
Arm/Group | IM20 Group | IM60 Group | Blank Control Group
Number analyzed (Participants) | 155 | 150 | 151
Participants | 27 | 44 | 0

ADVERSE EVENTS:
Description: The blank control group was not vaccinated with hepatitis B vaccine, so adverse reactions of hepatitis B vaccine were not collected and analyzed.
Arm/Group | IM20 Group | IM60 Group
All-Cause Mortality (participants affected / at risk) | 0/158 | 0/156
Serious Adverse Events (participants affected / at risk) | 0/158 | 0/156
Other Adverse Events (participants affected / at risk) | 12/158 | 11/156
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IM20 Group (N=158) | IM60 Group (N=156)
erytherma (Skin and subcutaneous tissue disorders) | 8 | 9
pain (Musculoskeletal and connective tissue disorders) | 10 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No